CLINICAL TRIAL: NCT05592444
Title: Different Strategies to Reduce Contrast Medium in Computed Tomography Pulmonary Angiography Using Spectral Detector CT
Brief Title: Strategies to Reduce Contrast Medium in Spectral CT Pulmonary Angiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Peter Maehre Lauritzen, Principal Investigator, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 142126
Record Dates: First submitted 2022-10-20; First posted 2022-10-24 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary Embolism; Spectral Detector CT; Contrast medium
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Intervention Model Description: Patients are randomly assigned to one of three injection methods: low concentration, low-volume and saline-dilution.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Acquired CT images are identical for all participants. The study arm is unknown to all, except the radiographers (radiology technicians) performing the examination.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low concentration (Experimental): Patients receive a contrast medium with an iodine concentration of 140 mg/ml. The volume is 1 ml/kg which result in a dose of 140 mg/kg.
  Maximal dose of contrast medium is 90 ml i.e. 12.6 g of iodine.
  Interventions: Diagnostic Test: Low iodine Spectral Detector CT Pulmonary Angiography
- Low volume (Experimental): Patients receive a contrast medium with an iodine concentration 350 of mg/ml. The volume is 0.4 ml/kg which result in a dose of 140 mg/kg.
  Maximal dose of contrast medium is 36 ml i.e. 12.6 g of iodine.
  Interventions: Diagnostic Test: Low iodine Spectral Detector CT Pulmonary Angiography
- Saline Dilution (Experimental): Patients receive a contrast medium with an iodine concentration of 350 mg/ml. The contrast medium is diluted 1:1 with saline.
  The injected volume is 0.8 ml/kg which result in a dose of 140 mg/kg. Maximal dose of contrast medium is 72 ml i.e. 12.6 g of iodine.
  Interventions: Diagnostic Test: Low iodine Spectral Detector CT Pulmonary Angiography

INTERVENTIONS:
Diagnostic Test: Low iodine Spectral Detector CT Pulmonary Angiography — Low iodine Spectral Detector CT Pulmonary Angiography

SUMMARY:
The purpose of this study is to assess the effect of three different strategies to inject at reduced volume of contrast medium in Computed Tomography Pulmonary Angiography (CTPA).

330 patients referred for CTPA are randomized to receive either a low-concentration, a low-volume or a saline-diluted injection.

Effects on the level and homogeneity of contrast enhancement are measured and compared between groups.

DETAILED DESCRIPTION:
Spectral detector CT facilitates large reductions in contrast medium in vascular CT examinations. To our knowledge, no studies have so far compared different strategies to inject this reduced contrast dose.

The purpose of this study is to assess the effect of three different strategies to inject at reduced volume of contrast medium in Computed Tomography Pulmonary Angiography (CTPA).

330 patients referred for clinically indicated CTPA are randomized to receive either a low-concentration, a low-volume or a saline-diluted injection. All patients receive the same amount of iodine (140 mg/kg).

Effects on the level and homogeneity of contrast enhancement, image noise, contrast-to-noise-ratio and signal-to-noise-ratio are measured in the CT images and the results are compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients and outpatients with kidney function (eGFR) allowing for safe administration of contrast dose (as calculated with the OmniVis calculator).
* Patients with clinical suspicion of disease of PE
* Referral to CTPA diagnosis, treatment planning or follow-up.
* Peripheral venous catheter (PVC) =/< 18 G

Exclusion Criteria:

* Contraindication to iodinated contrast medium
* Age < 18 years
* Lack of informed consent
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
Contrast enhancement (Vascular attenuation) | Measured on the CT images from the examination performed at enrollment
  Contrast enhancement measured as attenuation in the pulmonary artery Branches on the acquired CTPA examination

SECONDARY OUTCOMES:
Homogeneity of contrast enhancement (image noise) | Measured on the CT images from the examination performed at enrollment
  Homogeneity of contrast enhancement is measured as the standard deviation of attenuation in the pulmonary artery branches (equals image noise).
Contrast to noise ratio (CNR) | Measured on the CT images from the examination performed at enrollment
  CNR is measured as (Vascular attenuation - Muscular attenuation) / Image noise
Signal to noise ratio (SNR) | Measured on the CT images from the examination performed at enrollment
  SNR is measured as Vascular attenuation / Image noise

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Lauritzen, PhD, Principal Investigator — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, Lørenskog, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No